CLINICAL TRIAL: NCT01842568
Title: Vascular Events In Surgery patIents cOhort evaluatioN - Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Abbott Diagnostics Division (Industry)
Responsible Party: Principal Investigator, Andre Lamy, Professor and Cardiac Surgeon, Population Health Research Institute
Other Study IDs: VISION Cardiac Surgery
Record Dates: First submitted 2013-04-17; First posted 2013-04-29 (Estimated); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Vascular Death; Myocardial Infarction; Stroke; Cardiac Surgery
Keywords: Cardiac surgery; Troponin; Vascular events; Myocardial injury; Observational cohort study; Public health
MeSH Terms: conditions — Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Worldwide over 2 million adults (>30,000 Canadians) undergo heart surgery annually. Although heart surgery provides important survival benefits, it is associated with potential major complications such as death, stroke, and heart attack. There is promising evidence that measurement of heart injury markers after surgery will identify patients at risk of death or major complications.

This study will determine the current incidence of major complications in a representative sample of 15,000 contemporary adult patients undergoing heart surgery. Knowing the current burden of complications will inform clinicians, administrators, government and granting agencies about resources required to address the problem. This study will also establish the role of measuring heart injury markers to identify important heart injury after heart surgery and the proportion that would go undetected without routine heart injury marker monitoring. This information will facilitate further studies of timely interventions. In summary, the VISION Cardiac Surgery Study addresses fundamental questions that will have profound public health implications given the millions of adults worldwide who undergo heart surgery annually.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Patients who have undergone cardiac surgery. This includes coronary artery bypass grafting and all open heart procedures such as valvular repairs/replacement.

Exclusion Criteria:

1. Previously enrolled in the VISION Cardiac Surgery Study.
2. Patients who have undergone an isolated pericardial window, pericardiectomy, permanent pacemaker or defibrillator implantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have undergone cardiac surgery who are at least 18 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 15989 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2022-05 (Actual); Study Completion 2025-07 (Actual)

PRIMARY OUTCOMES:
All-cause mortality at 30-days after surgery | 30 days after surgery
  All-cause mortality at 30-days after surgery
Myocardial injuries that were not identified clinically during the first 5 days after surgery | 5 days after surgery
  Myocardial injuries that were not identified clinically during the first 5 days after surgery
Composite of vascular death, nonfatal myocardial infarction, nonfatal cardiac arrest, nonfatal stroke, and mechanical assist device | 30 days after surgery
  Major vascular complications at 30 days after surgery (i.e., a composite of vascular death, nonfatal myocardial infarction, nonfatal cardiac arrest, nonfatal stroke, and mechanical assist device)
Composite of vascular death, nonfatal myocardial infarction, nonfatal cardiac arrest, nonfatal stroke, and mechanical assist device | 1 year after surgery
  Major vascular complications at 1-year after surgery (i.e., a composite of vascular death, nonfatal myocardial infarction, nonfatal cardiac arrest, nonfatal stroke, and mechanical assist device)

SECONDARY OUTCOMES:
Composite of vascular death, nonfatal myocardial infarction, nonfatal stroke, and mechanical assist device | 30 days after surgery
  Major vascular complications at 30-days after surgery (i.e., a composite of vascular death, nonfatal myocardial infarction, nonfatal stroke, and mechanical assist device)
Total mortality | 30 days after surgery
  Total mortality
Total mortality | 1 year after surgery
  Total mortality
Vascular mortality | 30 days after surgery
  death due to vascular cause
Vascular mortality | 1 year after surgery
  death due to vascular cause
Myocardial infarction | 30 days after surgery
  Myocardial infarction
Myocardial infarction | 1 year after surgery
  Myocardial infarction
Non-fatal cardiac arrest | 30 days after surgery
  Non-fatal cardiac arrest
Non-fatal cardiac arrest | 1 year after surgery
  Non-fatal cardiac arrest
Stroke | 30 days after surgery
  Stroke
Stroke | 1 year after surgery
  Stroke
Implantation of mechanical assist device | 30 days after surgery
  Implantation of mechanical assist device
Implantation of mechanical assist device | 1 year after surgery
  Implantation of mechanical assist device
Cardiac transplant | 30 days after surgery
  Cardiac transplant
Cardiac transplant | 1 year after surgery
  Cardiac transplant
Repeat cardiac revascularization procedures | 30 days after surgery
  Repeat cardiac revascularization procedures
Repeat cardiac revascularization procedures | 1 year after surgery
  Repeat cardiac revascularization procedures
Congestive heart failure | 30 days after surgery
  Congestive heart failure
Congestive heart failure | 1 year after surgery
  Congestive heart failure
New atrial fibrillation | 30 days after surgery
  New clinically important atrial fibrillation
New atrial fibrillation | 1 year after surgery
  New clinically important atrial fibrillation
Pulmonary embolus | 30 days after surgery
  Pulmonary embolus
Pulmonary embolus | 1 year after surgery
  Pulmonary embolus
Deep venous thrombosis | 30 days after surgery
  Deep venous thrombosis
Deep venous thrombosis | 1 year after surgery
  Deep venous thrombosis
Major bleeding | 30 days after surgery
  Major bleeding
Major bleeding | 1 year after surgery
  Major bleeding
New dialysis | 30 days after surgery
  New dialysis
New dialysis | 1 year after surgery
  New dialysis
Infection | 30 days after surgery
  Infection (including sternal, sepsis, pneumonia)
Infection | 1 year after surgery
  Infection (including sternal, sepsis, pneumonia)
Re-hospitalization for a vascular reason | 30 days after surgery
  Re-hospitalization for a vascular reason
Re-hospitalization for a vascular reason | 1 year after surgery
  Re-hospitalization for a vascular reason
Chronic incisional pain | 30 days after surgery
  Chronic incisional pain
Chronic incisional pain | 1 year after surgery
  Chronic incisional pain
Frailty | 30 days after surgery
  Frailty assessed by PRISMA-7 questionnaire
Frailty | 1 year after surgery
  Frailty assessed by PRISMA-7 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: P.J. Devereaux, MD, PhD, Study Chair — McMaster University; Andre Lamy, MD, Principal Investigator — McMaster University; Richard Whitlock, MD, Principal Investigator — McMaster University
Locations (24):
- Ronald Reagan Medical Centre, UCLA, Los Angeles, California, United States
- Royal Prince Alfred Hospital, Sydney, New South Wales, Australia
- Brazil (3):
  - Hospital de Clínicas de Porto Alegre - HCPA, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia do RS, Porto Alegre, Rio Grande do Sul
  - INCOR, São Paulo
- Canada (3):
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
- First Teaching Hospital, Xinjiang, China
- Prince of Wales Hospital, Shatin, Hong Kong, SAR, Hong Kong
- Italy (3):
  - Santa Maria Hospital, GVM Care and Research, Bari
  - University of Bari "Aldo Moro", Bari
  - San Raffaele Scientific Institute, Milan
- Malaysia (2):
  - Institut Jantung Negara Sdn. Bhd., Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
- Department of Cardiovascular Surgery, Medical University of Gdansk, Gdansk, Poland
- Russia (2):
  - Federal State Budgetary Institution "Research Institute for Complex Issues of Cardiovascular Diseases", Kemerovo
  - Research Institute of Circulation Pathology, Novosibirsk
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- United Kingdom (5):
  - Essex Cardiothoracic Centre, Basildon and Thurrock University NHS Trust, Basildon, Essex
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, Lancashire
  - Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, Merseyside
  - BHF Centre of Cardiovascular Science, University of Edinburgh, Edinburgh
  - New Cross Hospital, Wolverhampton

REFERENCES:
- [Derived] Devereaux PJ, Lamy A, Chan MTV, Allard RV, Lomivorotov VV, Landoni G, Zheng H, Paparella D, McGillion MH, Belley-Cote EP, Parlow JL, Underwood MJ, Wang CY, Dvirnik N, Abubakirov M, Fominskiy E, Choi S, Fremes S, Monaco F, Urrutia G, Maestre M, Hajjar LA, Hillis GS, Mills NL, Margari V, Mills JD, Billing JS, Methangkool E, Polanczyk CA, Sant'Anna R, Shukevich D, Conen D, Kavsak PA, McQueen MJ, Brady K, Spence J, Le Manach Y, Mian R, Lee SF, Bangdiwala SI, Hussain S, Borges FK, Pettit S, Vincent J, Guyatt GH, Yusuf S, Alpert JS, White HD, Whitlock RP; VISION Cardiac Surgery Investigators. High-Sensitivity Troponin I after Cardiac Surgery and 30-Day Mortality. N Engl J Med. 2022 Mar 3;386(9):827-836. doi: 10.1056/NEJMoa2000803. PMID 35235725
- [Derived] Spence J, Bosch J, Chongsi E, Lee SF, Thabane L, Mendoza P, Belley-Cote E, Whitlock R, Brady K, McIntyre WF, Lamy A, Devereaux PJ. Standardized Assessment of Global activities in the Elderly scale in adult cardiac surgery patients. Br J Anaesth. 2021 Oct;127(4):539-546. doi: 10.1016/j.bja.2021.05.037. Epub 2021 Jul 28. PMID 34330417
- [Derived] McGillion MH, Henry S, Busse JW, Ouellette C, Katz J, Choiniere M, Lamy A, Whitlock R, Pettit S, Hare J, Gregus K, Brady K, Dvirnik N, Yang SS, Parlow J, Dumerton-Shore D, Gilron I, Buckley DN, Shanthanna H, Carroll SL, Coyte PC, Ebrahim S, Isaranuwatchai W, Guerriere DN, Hoch J, Khan J, MacDermid J, Martorella G, Victor JC, Watt-Watson J, Howard-Quijano K, Mahajan A, Chan MTV, Clarke H, Devereaux PJ. Examination of psychological risk factors for chronic pain following cardiac surgery: protocol for a prospective observational study. BMJ Open. 2019 Mar 1;9(2):e022995. doi: 10.1136/bmjopen-2018-022995. PMID 30826789
- [Derived] Ackland GL, Abbott TEF, Cain D, Edwards MR, Sultan P, Karmali SN, Fowler AJ, Whittle JR, MacDonald NJ, Reyes A, Paredes LG, Stephens RCM, Del Arroyo AG, Woldman S, Archbold RA, Wragg A, Kam E, Ahmad T, Khan AW, Niebrzegowska E, Pearse RM. Preoperative systemic inflammation and perioperative myocardial injury: prospective observational multicentre cohort study of patients undergoing non-cardiac surgery. Br J Anaesth. 2019 Feb;122(2):180-187. doi: 10.1016/j.bja.2018.09.002. Epub 2018 Oct 2. PMID 30686303